CLINICAL TRIAL: NCT03779425
Title: VR-Based Physical Therapy Pilot Study
Acronym: VR-PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: KairosXR (Other); AO North America (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D19021
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Extremity Fracture Lower

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Physical Therapy (Experimental): Participants will undergo a non-weight bearing knee range of motion virtual reality physical therapy session.
  Interventions: Other: Virtual Reality Physical Therapy

INTERVENTIONS:
Other: Virtual Reality Physical Therapy — Participants will undergo a non-weight bearing knee range of motion virtual reality physical therapy session.

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of using the virtual reality-based physical therapy platform in patients with extremity fracture.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Diagnosed with an operative fracture of the femur and/or tibia
* referred to physical therapy as standard of care

Exclusion Criteria:

* Injury Severity Score(ISS) > 18
* bilateral lower extremity injuries that preclude crutch ambulation
* associated spine fractures
* Glasgow Coma scale (GCS) < 15 at time of discharge
* major peripheral nerve injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Assessed directly after virtual reality physical therapy session
  Patient satisfaction with the virtual reality based physical therapy platform. Patient satisfaction will be assessed using a questionnaire created for this study.
Patient Preference | Assessed directly after virtual reality physical therapy session
  Patient preference for virtual reality-based physical therapy when compared to standard supervised office based physical therapy. Patient preference will be assessed using a questionnaire created for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States